CLINICAL TRIAL: NCT00818506
Title: Associations Between Depression and Cardiovascular Disease in Patients With Late Onset, Single Episode Major Depressive Disorder
Brief Title: Associations Between Depression and Cardiovascular Disease - a Study of Patients With Late Onset Depression
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Ministry of Science, Technology and Innovation, Denmark (Other Government); Vejle Hospital (Other); Danish National Research Foundation (Other); Aarhus University Hospital (Other); Augustinus Fonden (Other)
Responsible Party: Sponsor
Other Study IDs: CPF-TAD-1
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Depression; Major Depressive Disorder; Cardiovascular Disease; Coronary Artery Disease
Keywords: Depression; Major depressive disorder; Coronary artery disease; White Matter Hyperintensities; White Matter Lesions; Coronary artery calcification
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Late onset MDD: Patients with major depressive disorder between 50 and 70 years of age that did not suffer from depression before the age of 50.
- Controls: Healthy controls (matched for age, sex, and tobacco use status)

SUMMARY:
Studies show that depression is a risk factor for the development of coronary artery disease (CAD). Furthermore there is an increased occurrence of depression in patients with CAD. Among other mechanisms atherosclerosis is believed to play a central role regarding these notable associations between depression and CAD. Moreover, patients with late onset major depression have an increased number of small lesions found in the white matter of the brain, the so-called white matter lesions. The main goal of this project is to examine if CAD is associated with depression and/or white matter lesions. CAD is evaluated using coronary CT angiography. Depression is evaluated using a semi-structured diagnostic interview. White matter lesions are quantified using cerebral magnetic resonance.

ELIGIBILITY:
INCLUSION CRITERIA:

* Submitted to psychiatric hospital, district psychiatry or private psychiatrist because of major depressive disorder.
* Meets the criteria for Major Depressive Disorder, Single Episode as defined in the Diagnostic and Statistical Manual, fourth edition (DSM-IV) and the International Classification of Diseases (ICD-10).
* Age 50-70 years.
* Written informed consent.
* Caucasian.

EXCLUSION CRITERIA:

* Known, or anamnestic/objective signs of, organic brain disease.
* Organic, including symptomatic, mental disorders as (ICD-10: F00-F09).
* Dependence syndrome within the last 5 years (ICD-10: F1x.2) or current harmful use (ICD-10: F1x.1) of alcohol or other psychoactive substances.
* Schizophrenia, schizotypal and delusional disorders (ICD-10: F20-F29).
* Subject to force of law according to the danish law on psychiatry.
* Present risk of suicide.
* Previous cranial trauma resulting in unconsciousness for more than 2 minutes.
* Medical history of renal failure.
* Other conditions which contraindicate specific procedures in the project.
* Other conditions deemed to prevent the subject from completing the examination program.
* Does not want to participate.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatric treatment facilities (e.g. psychiatric hospital, private psychiatrist).
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-03; Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Poul Videbech, Professor, M.D., Dr.Med., Study Director — Center of Psychiatric Research, Aarhus University Hospital
Locations (1):
- Center of Psychiatric Research, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- See also: Center of Psychiatric Research, Aarhus University Hospital — http://psykiatriskforskning.dk/english/